CLINICAL TRIAL: NCT02135393
Title: Folic Acid Handling by the Human Gut: Implications for Food Fortification and Supplementation
Brief Title: Where is the Initial Site of Biotransformation of Folates in Humans?
Acronym: FOLTIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Quadram Institute Bioscience (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UK CRN 5085
Record Dates: First submitted 2014-05-08; First posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 13C5-folic acid or 13C5-6S-5-FormylTHF (Experimental): Physiological 500 nmol (220 µg folic acid equivalent) dose of dietary supplement 13C5-folic acid or 13C5-6S-5-FormylTHF given to subjects with in situ transjugular intrahepatic portosystemic stent at the time of routine venography patency check followed by regular portal venous sampling for 85 minutes at pre determined intervals and then physiological 500 nmol dose of 13C-6S-5-FormylTHF or 13C5-folic acid respectively at the next annual routine venography patency check followed by portal venous sampling for 85 minutes
  Interventions: Dietary Supplement: 13C5-folic acid or 13C5-6S-5-FormylTHF

INTERVENTIONS:
Dietary Supplement: 13C5-folic acid or 13C5-6S-5-FormylTHF — Subjects with an insitu transjugular intrahepatic porto systemic stent shunt assigned to receive either a physiological 500 nmol (220 µg folic acid equivalent) dose of 13C5-folic acid or 13C5-6S-5-FormylTHF at the time of routine shunt venography to check patency followed by portal venous sampling at pre defined time points for 85 minutes and then given 13C5-6S-5-FormylTHF ator 13C5-folic acid at their next annual venography patency check with portal venous sampling at pre defined time points for 85 minutes

SUMMARY:
The aim of this study is to test the assumption that, in humans, folic acid, a dietary supplement is biotransformed (reduced and methylated) to the natural circulating plasma folate 6S-5Methyltetrahydrofolic acid (5-MTHF) in the intestinal mucosa.

DETAILED DESCRIPTION:
Current thinking, based mainly on rodent studies, is that physiological doses of folic acid (pteroylmonoglutamic acid), like dietary vitamin folates, are biotransformed in the intestinal mucosa and transferred to the portal vein as the natural circulating plasma folate, 5-methyltetrahydrofolic acid (5-MTHF), before entering the liver and the wider systemic blood supply.

Study design:Open labelled study that samples portal and peripheral veins for labelled folate concentrations following oral ingestion with physiological doses of dietary supplements stable-isotope-labelled folic acid, or, the reduced folate, 5-formyltetrahydrofolic acid (5-FormylTHF). The study was performed in subjects with a Transjugular Intrahepatic Porto Systemic Shunt (TIPSS) in situ at the time of a routine annual patency check to allow blood samples to be taken from the portal vein. The aim of this study is to test the assumption that, in humans, folic acid is biotransformed (reduced and methylated) to 5-MTHF in the intestinal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Stable, synthetic liver function without recent evidence of decompensation (defined as liver function inadequacy or active complications of portal hypertension)
* Abstinent from alcohol
* Free from malignant disease
* Normal gut permeability (as assessed by the lactulose/mannitol test)
* Patent TIPSS on their last surveillance

Exclusion Criteria:

* Taking Vitamin B supplements
* Taking Folic Acid supplementation
* Unable to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The percentage of folate in un-modified and modified form in the portal vein for each of the different oral folate dosing formulations | 85 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David E Jones, PhD FRCP, Principal Investigator — Newcastle University
Locations (2):
- United Kingdom (2):
  - Freeman Hospital, Newcastle upon Tyne, Tyneside
  - Institute of Food Research, Norwich

REFERENCES:
- [Derived] Patanwala I, King MJ, Barrett DA, Rose J, Jackson R, Hudson M, Philo M, Dainty JR, Wright AJ, Finglas PM, Jones DE. Folic acid handling by the human gut: implications for food fortification and supplementation. Am J Clin Nutr. 2014 Aug;100(2):593-9. doi: 10.3945/ajcn.113.080507. Epub 2014 Jun 18. PMID 24944062